CLINICAL TRIAL: NCT03383796
Title: Randomized Clinical Trial Comparing Three Dimension Laparoscopic and Open Surgery for Perihiliar Cholangiocarcinoma
Brief Title: Comparing Three Dimension Laparoscopic Versus Open Surgery for Perihiliar Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Clinical professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJDBPS02
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cholangiocarcinoma, Perihilar; Surgery
Keywords: Cholangiocarcinoma perihilar; three dimension laparoscopic
MeSH Terms: conditions — Klatskin Tumor | interventions — 6-propylchromone-2-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D approach (Experimental): Three dimensional laparoscopic resection for pCCA
  Interventions: Procedure: Three dimensional laparoscopic resection for pCCA
- open approach (Experimental): Open resection for pCCA
  Interventions: Procedure: Open resection for pCCA

INTERVENTIONS:
Procedure: Three dimensional laparoscopic resection for pCCA — Three dimensional laparoscopic resection for pCCA
  Arms: 3D approach
Procedure: Open resection for pCCA — Open resection for pCCA
  Arms: open approach

SUMMARY:
Cholangiocarcinoma (CCA) is the most common biliary tract malignancy and the second most common primary hepatic malignancy. The prognosis of CCA is dismal. Surgery is the only potentially curative treatment, but the majority of patients present with advanced stage disease, and recurrence after resection is common. It is classified into intrahepatic (iCCA), perihilar (pCCA), and distal (dCCA) subtypes. Among all, pCCA is the most common subtype.

This is a prospective, randomized, controlled multicenter trial with two treatment arms, three dimension laparoscopic approach versus open approach. The trial hypothesis is that three dimension laparoscopic surgery has advantages in postoperative recoveries and be equivalent in operation time, oncological results and long-term follow-up compared with open counterpart. The duration of the entire trial is two years including prearrangement, follow-up and analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven pCCA.
2. Highly presumed perihlar bile duct malignancy with difficulties to obtain histological evidence.
3. Preoperative staging work up performed by upper abdomen enhanced CT scan.
4. The subject understands the nature of this trial and willing to comply.
5. Ability to provide written informed consent.
6. Patients treated with curative intent in accordance to international guidelines

Exclusion Criteria:

1. Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs.
2. Subjects undergoing any part for hepatectomy.
3. Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score >4.
4. Synchronous malignancy in other organs.
5. Palliative surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 months
  Mortality was defined as any death that occurred in the 30 days after surgery or during the hospital stay.
Length of Stay | 24 months
  Length of stay was defined as the postoperative time interval in days.
R0 Resection Rate | 24 months
  Negative margin rate.
Bile leakage | 24 months
  The drain bilirubin was monitored after surgery, any elevation for the bilirubin level or the diagnostic puncture proved bile fluid in abdominal cavity.
TNM Staging | 24 months
  According to AJCC guideline, each patients TNM staging were recorded.
Complication rate | 24 months
  Complication Rate Measure Description Any complication mentioned in the protocol should be carefully record and analyzed, including postoperative hemorrhage, postoperative pancreatic fistula, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided